CLINICAL TRIAL: NCT06026111
Title: Preliminary Efficacy of Different Exercise Training During Immunotherapy in Patients With Lung Cancer: The ENHANCE Trial
Acronym: ENHANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-247
Record Dates: First submitted 2023-08-10; First posted 2023-09-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Intensity Interval Training (HIIT) (Experimental): Patients in the HIIT group will perform alternating vigorous-intensity and recovery aerobic exercise intervals on a provided home stationary bike. The HIIT protocol consists of alternating a high-intensity exercise phase (1 min at 65-90% of workload corresponding to VO2peak) and a recovery phase (1 min at 30%), and the high-intensity and recovery intervals will be repeated 5-10 times in each session.
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)
- Moderate-Intensity Continuous Training (MICT) (Experimental): The MICT group will perform an aerobic exercise at a continuous intensity in each session on a stationary bike. Similar to HIIT, the intensity will be progressed (47.5-60%). The total work of MICT is equalized with HIIT for training volume and frequency to compare the differences exerted from different intensities and energy expenditure.
  Interventions: Behavioral: Moderate-Intensity Continuous Training (MICT)
- Usual Care (UC) (No Intervention): Participants will be asked to maintain their baseline exercise behavior and will be offered to participate in the HIIT exercise program upon the completion of post-intervention assessments after the initial 12 weeks.

INTERVENTIONS:
Behavioral: High-Intensity Interval Training (HIIT) — Home-based, virtually supervised, aerobic exercise intervention at a high intensity in an interval fashion.
  Arms: High-Intensity Interval Training (HIIT)
Behavioral: Moderate-Intensity Continuous Training (MICT) — Home-based, virtually supervised, aerobic exercise intervention at a moderate intensity in a continuous fashion.
  Arms: Moderate-Intensity Continuous Training (MICT)

SUMMARY:
The purpose of this study is to examine the feasibility and effects of 12-week exercise training at different intensities among individuals with advanced lung cancer receiving immune checkpoint inhibitors.

The names of the study interventions involved in this study are:

DETAILED DESCRIPTION:
This single-center, two-armed, pilot randomized controlled research study will assess feasibility and compare immune activities, cardiorespiratory fitness, physical function, and immunotherapy-related adverse events, and patient-reported outcomes between three groups - high-intensity exercise, moderate-intensity exercise, and usual care.

Participants in this study will be randomly assigned to one of three groups:

* High-intensity interval training (HIIT)
* Moderate-intensity continuous training (MICT)
* Usual care (UC) The HIIT and the MICT groups will receive virtually supervised home-based exercise training three sessions per week for 12 weeks. The UC group will be asked not to change their baseline exercise behavior and will be offered to receive one of the exercise programs at the end of the initial 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically diagnosed with advanced non-small cell lung cancer (NSCLC).
* Having been receiving anti-PD-1 or anti-PD-L1 antibodies (i.e., single agent or combination) for at least one month with a plan to continue for at least 12 weeks prospectively at the time of recruitment.
* Medical clearance to perform exercise intervention and testing by their treating oncologist.
* No uncontrolled medical conditions that could be exacerbated with exercise (e.g., uncontrolled hypertension or diabetes).
* Ability to communicate and complete written forms in English.
* Participate in less than or equal to 60 minutes of moderate-to-vigorous aerobic exercise per week over the past month.
* Ability to understand and the willingness to sign informed consent prior to any study-related procedures.
* Willing to travel to DFCI for necessary data collection.

Exclusion Criteria:

* Participate in more than 60 minutes of moderate-to-vigorous aerobic exercise per week over the past month. This study targets insufficiently active persons to assess the effect of the described exercise intervention, where additional exercise done regularly will contaminate the intervention outcomes.
* Unstable comorbidities that prevent participation in moderate-to-vigorous intensity exercise. Patients with unstable comorbidities may develop unexpected adverse events from exercise. For the purpose of patients' safety, as well as because part of this study involves remote, home-based exercise where close supervision is not possible, patients with unstable medical conditions are excluded.
* Subjects who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Development of second malignancy (except for basal cell carcinoma or squamous cell carcinoma of the skin) that requires concurrent treatment, which would interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants completing the exercise intervention sessions | Up to 14 weeks
  The primary outcome is feasibility and will be assessed by the proportion of enrolled participants completing the exercise intervention sessions with >/=70% completion considered feasible.

SECONDARY OUTCOMES:
Neutrophil-lymphocyte ratio (NLR) | Baseline (Week 1) and post-intervention (Week 14)
  Neutrophil-lymphocyte ratio (NLR) will be assessed as a systemic immune marker as well as a prognostic marker of immunotherapy. Mononuclear lymphocyte phenotypes will be conducted in the Immune Assessment Laboratory. Immunofluorescence assays in whole blood will identify the counts of neutrophils and lymphocytes. Fasting blood will be taken in the morning following an overnight fast. Two 10.0 mL EDTA tubes will be collected and one spun for 10 minutes at 2860rpm within one hour of collection and 1.0mL of plasma will be transferred to a secondary tube to cryovials. Samples will be stored or shipped frozen at -70°C. Samples will be centrifuged, stored at -80°C, and batch-analyzed after post-intervention assessments.
Cardiopulmonary Fitness | Baseline (Week 1) and post-intervention (Week 14)
  Cardiorespiratory fitness will be assessed as VO2peak by a graded maximal cycle exercise stress test. VO2peak is defined as the highest values of oxygen uptake averaged among every 15-second interval during the test. VO2peak will be reported in both relative (ml·kg-1·min-1) and absolute (L/min) terms.
Muscular Strength | Baseline (Week 1) and post-intervention (Week 14)
  Muscular strength will be measured as 1-repetition maximum (RM) (i.e., the greatest resistance that can be moved through the full range of motion), which has been the standard for strength assessments. 1-RM values will be estimated from 10-RM using validated equations on 12 exercises including the ten exercises utilized in the prescription not performed on machines.
Short Physical Performance Battery | Baseline (Week 1) and post-intervention (Week 14)
  Physical function will be assessed by the Short Physical Performance Battery (SPPB), which includes the following 3 lower extremity measures completed in the following order. Timed balance (seconds): Balance will be assessed under 3 conditions (side-by-side, semi-tandem, and tandem stands). Gait speed (seconds): Gait speed will be assessed over a 4-meter flat surface distance. The participant will be asked to complete 2 attempts of this test. Time will be recorded using an electronic timing system. Chair stand (seconds): Chair stand will be performed under 2 conditions: a) subjects will perform a single chair stand; b) subjects will be asked to perform 5 repeated chair stands as quickly as possible; time to completion will be recorded.
Patient Reported Outcomes - Health-related quality of life | Baseline (Week 1) and post-intervention (Week 14)
  quality of life will be assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ)-C30.
Patient Reported Outcomes - Lung-cancer related quality of life | Baseline (Week 1) and post-intervention (Week 14)
  Lung-cancer related quality of life will be assessed by the European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-Lung Cancer (EORTC-QLQ-LC)-29.
Patient Reported Outcomes - Immunotherapy Symptoms | Baseline (Week 1) and post-intervention (Week 14)
  Immunotherapy symptoms will be assessed by the MD Anderson Symptom Inventory (MDASI) Immunotherapy early-phase trials (EPT).
Patient Reported Outcomes - Anxiety and Depression | Baseline (Week 1) and post-intervention (Week 14)
  Anxiety and Depression will be assess using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, divided into two 7-item subscales (anxiety and depression). The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence) and the total score is out of 42 (21 per subscale).
Patient Reported Outcomes - Sleep Quality | Baseline (Week 1) and post-intervention (Week 14)
  Sleep will be assessed using the Pittsburg Sleep Quality Index (PSQI).

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu